CLINICAL TRIAL: NCT04325087
Title: Reduction of Trauma-induced Intrusions and Amygdala Hyperreactivity Via Non-invasive Brain Stimulation
Acronym: COOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor Rene Hurlemann, M.Sc., M.D., Ph.D., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: COOL
Record Dates: First submitted 2020-02-28; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Intrusive Thoughts; Post Traumatic Stress Disorder
Keywords: Amygdala; fMRI; Intrusive Thoughts; Post Traumatic Stress Disorder; TMS
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants receive either three sessions of iTBS over the dorsolateral prefrontal cortex or three sessions of a placebo stimulation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active iTBS (Experimental): Active stimulation of the dlPFC directly after trauma exposure and on the following two days
  Interventions: Device: iTBS
- Placebo iTBS (Placebo Comparator): Same procedure as in the active stimulation group but with a placebo stimulation imitating the sensation of a real iTBS protocol.
  Interventions: Device: Placebo iTBS

INTERVENTIONS:
Device: iTBS — Administration of an iTBS protocol over the dlPFC
  Arms: Active iTBS
Device: Placebo iTBS — Administration of a placebo TMS protocol over the dlPFC
  Arms: Placebo iTBS

SUMMARY:
The study will focus on the modulation of intrusive memories via functional magnetic resonance imaging (fMRI)-guided repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex (dlPFC) directly after exposure to a traumatic video.

DETAILED DESCRIPTION:
Traumatic experiences can lead to posttraumatic stress disorder (PTSD) with clinical manifestations including intrusions, avoidance behavior, and hyperarousal. Unlike most other psychological disorders, a PTSD diagnosis requires a clearly identifiable inciting event. As such, preventive interventions in recently traumatized individuals seem promising.

In this randomized, placebo-controlled study the investigators explore the potential of individualized transcranial magnetic stimulation (TMS) to reduce trauma-induced intrusive thoughts by altering functional connectivity between the dorsolateral prefrontal cortex (dlPFC) and amygdala. Subjects will undergo a functional magnetic resonance imaging (fMRI) session consisting of a resting state scan, an emotion recognition task and an anatomical scan at the beginning of the study (day 1). Resting state data will be used to determine individualized TMS targets for every subject, depending on functional connectivity between the dlPFC and amygdala. Subsequently, the analogue trauma model will be used to induce intrusions in healthy subjects. Subjects will be confronted with a video clip from the movie "Irreversible" and they will complete online questionnaires in the following three days to measure intrusive thoughts, trauma disclosure (i.e. duration of conversations about the aversive movie) and sleeping quality. Intermittent theta-burst stimulation (iTBS) will be administered directly after the video clip and on the following two days (day 2-4). Cognitive tasks will be applied before and after iTBS sessions to examine short-term effects of iTBS on a behavioral level. Finally, subjects will undergo a second fMRI session similar to the first one, to probe iTBS-induced changes in functional connectivity and emotional processing (day 5).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* current psychiatric illness
* current psychiatric medication or psychotherapy
* past PTSD diagnosis
* MRI contraindication (e.g. metal in body, claustrophobia)
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Number and quality of intrusive thoughts | Three days after trauma exposure
  Sum and stress ratings of intrusive thoughts measured on three consecutive days after trauma exposure by an online questionnaire.
Changes in resting state functional connectivity | 10-minutes resting state fMRI scans before and after three sessions of TMS treatment
  Functional connectivity data will be assessed by two 10-minutes resting state fMRI scans before and after three sessions of TMS treatment over the course of three days. The resting state fMRI analysis will focus on changes in functional connectivity between regions-of-interest (ROIs) associated with intrusive memories (prefrontal cortex, amygdala, precuneus, insula, hippocampus, cingulate cortex). Changes in functional connectivity between the first and second fMRI sessions will be computed on the first level and independent t-tests will be used to compare the verum and sham TMS groups.
Changes in neural response to an emotion recognition task | 15-minutes emotional face matching fMRI task before and after three sessions of TMS treatment
  Changes between the first and second fMRI session in the blood-oxygen-level-dependent (BOLD) signal in response to happy, fearful and neutral faces as well as houses will be compared between the experimental groups. Analysis will focus on anatomically defined regions-of-interest (ROI) associated with emotion processing (i.e. amygdala, prefrontal cortex, insula, striatal areas). Changes in the neural response and functional connectivity between the first and second fMRI sessions will be computed on the first level and independent t-tests will be used to compare the verum and sham TMS groups. For analyses of fMRI data, standard procedures of the software SPM12 will be used.

SECONDARY OUTCOMES:
Changes in executive functioning (One Touch Stockings of Cambridge) and attention (Rapid Visual Information Processing) during iTBS treatment | 15-minutes cognitive tasks pre/post first iTBS and pre/post last iTBS treatment
  Cognitive tasks conducted with the CanTab software will be used to measure executive functioning (One Touch Stockings of Cambridge) and attention (Rapid Visual Information Processing) on four different time points during the treatment (pre/post first iTBS, pre/post last iTBS). Changes in executive functioning and attention will be tested as moderator variables of other TMS effects.
Trauma disclosure | Three days after trauma exposure
  Trauma disclosure will be measured by online questionnaires on days 2-4. Subjects will be asked to report the number and duration (in minutes) of conversations about the video. Furthermore, subjects have to report to who they talked with about the video. Trauma disclosure will be tested as a moderator variable of TMS effects.
Changes in electrodermal responses to the trauma video | 5 minutes before and during the trauma video
  Electrodermal responses will be recorded by a BioNomadix System (BIOPAC Systems Inc., Santa Barbara, USA) during a 5-minutes baseline before the start of the trauma video and during the trauma video with two electrodes attached to palm of the right hand.
Respiratory changes in response to the trauma video | 5 minutes before and during the trauma video
  Respiratory rate will be recorded by a BioNomadix System (BIOPAC Systems Inc., Santa Barbara, USA) during a 5-minutes baseline before the start of the trauma video and during the trauma video with belt attached to the subject's chest. Data will be analyzed for changes in breathing frequency and amplitude in response to the trauma video.
Heart rate changes in response to the trauma video | 5 minutes before and during the trauma video
  Heart rate will be recorded by a BioNomadix System (BIOPAC Systems Inc., Santa Barbara, USA) during a 5-minutes baseline before the start of the trauma video and during the trauma video.
Changes in positive and and negative affect in response to the trauma video | 10 minutes before and 10 minutes after trauma exposure
  Changes in positive and negative affect will be measured by the PANAS (Positive and Negative Affect Schedule) questionnaire 10 minutes before and 10 minutes after trauma exposure. The PANAS questionnaire consists of two subscale: 1. positive affect (minimum rating = 5, maximum rating = 50), 2. negative affect (minimum rating = 5, maximum rating = 50).
Changes in anxiety in response to the trauma video | 10 minutes before and 10 minutes after trauma exposure
  Changes in anxiety will be measured by the STAI-Trait (State-Trait Anxiety Inventory) questionnaire immediately 10 minutes before and 10 minutes after trauma exposure.(minimum rating = 20, maximum rating = 80, higher values indicate more state anxiety).
Dissociative symptoms after trauma exposure | 10 minutes after trauma exposure
  Dissociative symptoms after the trauma video will be measured by questionnaires (Dissociation-Tension-Scale acute) and tested as a moderator variable of TMS effects. Subjects score between 0 and 9, with higher values indicating more dissociative symptoms.
Childhood maltreatment | Before first fMRI scan
  The Childhood Trauma Questionnaire (CTQ) will be used to measure childhood maltreatment. The scale ranges between 5 and 100 points and higher scores indicate higher childhood maltreatment. CTQ scores will be tested as moderator variable of TMS effects.
Sleep quality: visual analog scales | Three days after trauma exposure
  Sleep quality (delay in sleep onset, calmness, depth of sleep, nightmares, nightly awakenings) will be measured with visual analog scales from 0 to 100. Higher scores represent poor sleep quality.
Delayed discounting task | Before and three days after trauma exposure
  To test changes in PFC-associated control of impulsive preferences, subjects will perform a delayed discounting paradigm. Participants will be asked to choose between small immediate rewards and larger later rewards. This task will be conducted twice (before and after the iTBS sessions).
Food craving task | Before and three days after trauma exposure
  Food craving will be measured twice (before and after the iTBS sessions). Participants will be confronted with pictures of candy and dessert in two types of trials. In "NOW" trials, participants will be instructed to consider the immediate consequence of consuming the pictured food, while "LATER" trials will direct participants to think about the long-term consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc, MD, PhD, Principal Investigator — University of Oldenburg
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuromodulation of Emotion (NEMO) research group — http://renehurlemann.squarespace.com/welcome/